CLINICAL TRIAL: NCT00456586
Title: A 12-Week, Double-Blind, Placebo-Controlled, Randomized, Multicenter Study of the Efficacy of 40 mg/Day KW-6002 as Treatment for Parkinson's Disease in Patients With Motor Response Complications on Levodopa/Carbidopa Therapy
Brief Title: 12-Week, Double-Blind, Placebo-Controlled, Randomized Study of the Efficacy of 40 mg/Day KW-6002 in Parkinson's Disease Patients on Levodopa/Carbidopa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6002-US-005
Record Dates: First submitted 2007-04-03; First posted 2007-04-05 (Estimated); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Levodopa therapy; End of dose wearing off; Off time
MeSH Terms: conditions — Parkinson Disease | interventions — istradefylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: KW-6002 (istradefylline)

SUMMARY:
12-week, double-blind, placebo-controlled, multicenter, randomized study designed to evaluate the safety and efficacy of 40 mg/day istradefylline compared with placebo in subjects with OFF phenomena advanced PD who were treated with levodopa/carbidopa.

DETAILED DESCRIPTION:
A 12-week, double-blind, placebo-controlled, multicenter, randomized study designed to evaluate the safety and efficacy of 40 mg/day istradefylline compared with placebo in subjects with OFF phenomena advanced PD who were treated with levodopa/carbidopa.

ELIGIBILITY:
Inclusion Criteria:

1. United Kingdom Parkinson's Disease Society brain bank diagnostic criteria (step 1 and 2).
2. Modified Hoehn and Yahr Scale II-IV in the OFF state.
3. Treated with levodopa/carbidopa for 1 year with a stable regimen for 4 weeks prior to randomization.
4. Taking at least 4 doses of levodopa (3 doses if at least 2 doses containing slow release formulation) per day with predictable end of dose wearing off.
5. Successfully completed Parkinson's disease patient diary training with at least 120 minutes of OFF time per day.
6. Stable regimen of other antiparkinson's disease medications for at least 4 weeks prior to randomization.
7. At least 30 years of age and able to give written informed consent.

Exclusion Criteria:

1. Treatment with liquid levodopa/carbodopa within 4 weeks of randomization.
2. Treatment with MAO inhibitors except selegiline.
3. Treatment with centrally acting dopamine antagonists within 3 months (6 months for depot preparations), e.g., antipsychotic neuroleptics, metoclopramide, buspirone, amoxapine.
4. Neurosurgical surgery for Parkinson's disease.
5. Atypical parkinsonism or secondary parkinsonism variants.
6. Diagnosis of cancer or evidence of continued cancer within 5 years of enrollment or clinically significant illness of any organ system (e.g., ALT or AST > 1.5 times the upper limit of normal).
7. Mini-Mental Status Examination score of 25 or less.
8. History of drug or alcohol abuse or dependence within 2 years.
9. History of psychotic illness or seizures.
10. Current clinically relevant depression disorder.
11. History of neuroleptic malignant syndrome.
12. Pregnant or lactating females. Women of child-bearing potential must use reliable method of contraception.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2002-04; Primary Completion 2003-05 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of 40 mg/day istradefylline for reducing OFF time in subjects with Parkinson's disease (PD) treated with levodopa/carbidopa.

SECONDARY OUTCOMES:
To establish the efficacy of 40 mg/day istradefylline for reducing motor symptoms and improving activities of daily living (ADL) in subjects with advanced PD treated with levodopa/carbidopa.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sussman, MD, Study Director — Kyowa Kirin, Inc.
Locations (1):
- Contact Kyowa Pharmacuetical Inc., Princeton, New Jersey, United States